CLINICAL TRIAL: NCT04194840
Title: Pilot Study to Develop a Transplant Wellness Clinic for Elderly or High Risk Patients Undergoing Blood and Marrow Transplantation
Brief Title: Transplant Wellness Clinic for Elderly or High Risk Patients Undergoing BMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE9Z19
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Stem Cell Transplant Complications; Myeloma; Lymphoma; Allogeneic and Autologous Stem Cell Transplant
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma | interventions — Mental Status and Dementia Tests; Restraint, Physical; Medication Review; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transplant Wellness Clinic (Experimental): * Physical therapy consult
  * Intake vitals
  * CARG online survey, mental status exam
  * Medication review
  * Nutrition survey
  * Social work: available on prn basis (as-needed)
  * Exit survey
  Recommendations made and given to the participant and sent to the referring MD. Participant receives post clinic phone call before transplant. Referring MD receives questionnaires. Data collected depending on if participant moved forward with transplant
  Interventions: Other: physical therapy consult; Other: Cognitive Assessment; Other: Cancer Aging Research Group (CARG) assessment; Other: Medication Review; Other: Nutrition assessment; Other: Laboratory studies; Other: Patient satisfaction questionnaire; Other: Physician Questionnaire; Other: Patient follow-up questionnaire

INTERVENTIONS:
Other: physical therapy consult — Physical therapy consult to assess physical functioning on a separate office visit prior to attending the Transplant Wellness Clinic. Full evaluation that incorporates several tools to measure the risk of falling and to assess mobility and strength
Other: Cognitive Assessment — Montreal cognitive assessment (MoCA) and the Blessed Orientation-Memory-Concentration Test (BOMC)
Other: Cancer Aging Research Group (CARG) assessment — CARG assessment - utilized to capture information about a participant's medical history as well as functional, cognitive, and psychosocial status
Other: Medication Review — Medication Review via Beers Assessment
Other: Nutrition assessment — Nutrition assessment Via Mini Nutrition Assessment (MNA)
Other: Laboratory studies — Laboratory studies including urine toxicology screen, C-reactive protein, albumin, pre-albumin, vitamin D
Other: Patient satisfaction questionnaire — Patient satisfaction questionnaire
Other: Physician Questionnaire — Physician Questionnaire:
  Questionnaire to learn about physician satisfaction with information received from reports and participant questionnaires.
Other: Patient follow-up questionnaire — Patient follow-up questionnaire:
  Questionnaire to learn more about participant opinions concerning the clinic and the quality of care received during visits with specialists

SUMMARY:
As the average age of individuals undergoing stem cell transplant continues to increase, challenges associated with balancing the side effects of cancer treatments while also managing other medical conditions develop. Studies have shown these individuals develop more treatment related side effects and take longer to leave the hospital due to complications. The purpose of this study is to develop a multiple provider clinic that will help identify any additional needs in the more complicated and generally older transplant patient population. If needed, this clinic will recommend interventions or referrals to the appropriate specialties to the participant and the transplant physician for the participant before your transplant procedure. Examples of potential areas of improvement include a course of physical therapy, nutritional supplements, or modifications of medications, among others with the goal to make your transplant safer and to decrease length of time in the hospital.

DETAILED DESCRIPTION:
This is a supportive interventional study to assess frailty in at risk geriatric cancer patients undergoing stem cell transplant and to determine if specific interventions are feasible and will improve overall outcomes.

A total of 20 participants will be enrolled in this study with the first 10 participants limited to myeloma or lymphoma patients who meet eligibility criteria and are candidates for autologous transplantation. The second 10 participants enrolled will be either allogeneic or autologous stem cell transplant candidates who meet eligibility criteria.

The objectives of this study are as follows:

* To pilot a comprehensive multidisciplinary geriatric assessment clinic.
* To determine whether a comprehensive geriatric assessment (outside of physical therapy assessment) can be performed in a time efficient manner. The goal is to complete all questionnaires and the multidisciplinary assessments in <90 minutes.
* To assess participant and physician satisfaction
* To determine if interventions recommended in the clinic are achievable for each participant
* Examples of interventions could include, medication changes, management of depression, dietary modifications, physical therapy three times a week, etc.
* To determine if participation in the transplant wellness clinic reduces length of stay and readmission rate compared to historical controls at our institution

ELIGIBILITY:
Inclusion Criteria:

* Deemed candidate for autologous or allogeneic transplantation by their Stem Cell Transplant Attending Physician
* Stem cell transplant candidates > 60 years
* Younger patients with age adjusted HCT- CMI> 4
* Outpatient at time of enrollment.
* Must have at a minimum 4 weeks and a maximum of 12 weeks before anticipated start of transplant procedures, ie initiation of preparation regimen or beginning of peripheral stem cell mobilization
* Must have transportation to outpatient appointments
* Must be able to read and understand English to complete the required questionnaires Must be able to read and understand protocol consent

Exclusion Criteria:

- Those who are not felt to be candidates for autologous or allogeneic stem cell transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Time to complete geriatric assessment clinic | at time of assessment (an average of 90 minutes)
  Time to complete geriatric assessment clinic will be collected. Feasibility will be defined if 7 or more of the first 10 patients are able to complete the geriatric assessment clinic in under 90 minutes.
Patient satisfaction as determined by "patient follow-up quesitonnaire" | at time of assessment (less than 1 hour)
  Analysis of patient and physician questionnaires will be tabulated and results reported in a descriptive fashion
Physician satisfaction as determined by "physician questionnaire" | at time of assessment (less than 1 hour)
  Analysis of patient and physician questionnaires will be tabulated and results reported in a descriptive fashion
Length of transplant stay in days | Assessed up to 6 months after transplant
  Length of transplant stay will be collected for all participants and compared to historical controls of similar age
Readmission rates | Up to 100 days after transplant
  Readmission rates in the first 100 days post-transplant will be collected and compared to historical controls using Chi-square test

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Baer, APRN, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center; Brenda H Cooper, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Trial does not meet criteria for IPD sharing